CLINICAL TRIAL: NCT06705608
Title: Fingolimod and Risk of Skin Cancer Among Individuals with Multiple Sclerosis: a Population-based Cohort Study
Brief Title: Examining the Risk of Skin Cancer in Multiple Sclerosis Patients Using Fingolimod: a Population-Based Study
Acronym: MS; FTY720
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jacquelyn Cragg, Assistant Professor in the Faculty of Pharmaceutical Sciences, UBC, University of British Columbia
Other Study IDs: H24-03199
Record Dates: First submitted 2024-11-20; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis; Skin Cancer; Skin Cancer Melanoma; Skin Cancers - Basal Cell Carcinoma; Skin Cancer, Squamous Cell; Multiple Sclerosis (MS) - Relapsing-remitting
Keywords: multiple sclerosis and skin cancer; fingolimod; disease modifying therapy; FTY720; fingolimod and skin cancer
MeSH Terms: conditions — Multiple Sclerosis; Skin Neoplasms; Melanoma; Carcinoma, Basal Cell; Multiple Sclerosis, Relapsing-Remitting | interventions — Fingolimod Hydrochloride; Natalizumab; Dimethyl Fumarate; Alemtuzumab; teriflunomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients with multiple sclerosis: Adult participants with Multiple Sclerosis (MS), identified through a validated case definition, were observed in this retrospective cohort study. This case definition requires an individual to have at least three health care encounters (any combination of inpatient encounters, outpatient encounter, or disease-modifying-therapy (DMT) dispensation) for MS in a 1-year window. In this study, administrative claims data of participants between 2003 to 2020 were evaluated. The lower bound of this time period was selected based on data availability for the main drugs of interest. MS patients who initiated treatment with fingolimod or the active comparator drugs were identified to compare the incidence of skin cancer.
  Interventions: Drug: Fingolimod; Drug: Natalizumab; Drug: Dimethyl fumarate (DMF); Drug: Alemtuzumab; Drug: Teriflunomide

INTERVENTIONS:
Drug: Fingolimod — patients who received fingolimod for treating RRMS
Drug: Natalizumab — patients who received natalizumab for treating RRMS (active comparator)
Drug: Dimethyl fumarate (DMF) — patients who received dimethyl fumarate for treating RRMS (active comparator)
Drug: Alemtuzumab — patients who received alemtuzumab for treating RRMS (active comparator)
Drug: Teriflunomide — patients who received teriflunomide for treating RRMS (active comparator)

SUMMARY:
The goal of this retrospective observational study is to investigate the long-term safety of Fingolimod in individuals with Multiple Sclerosis (MS), specifically focusing on the risk of developing skin cancer. The main question it aims to answer is:

• Does the use of Fingolimod increase the incidence of skin cancer in individuals with MS compared to those using other disease-modifying therapies? Participants who are new users of Fingolimod or other active comparators as part of their regular medical care for MS will be included in this study. Researchers will use advanced causal inference techniques to analyze healthcare data and compare the incidence of skin cancer between these groups.

ELIGIBILITY:
Inclusion Criteria:

* Identified MS cohort with hospital/physician and prescription claims classified according to the international classification of disease codes and drug identification numbers respectively, using a validated case definition. This case definition requires an individual to have at least three health care encounters (any combination of inpatient encounter, outpatient encounter, or DMT dispensation) for MS in a 1-year window
* MS patients who initiated and used fingolimod, natalizumab, alemtuzumab, dimethyl fumarate, or teriflunomide as monotherapy following MS identification.

Exclusion Criteria:

* Pediatric (<18 years old) MS cases.
* MS cases with less than three years of baseline data before the first drug dispensation.
* MS cases with skin cancer in the three-year baseline period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with MS at age 18 or older who received fingolimod, natalizumab, alemtuzumab, DMF, or teriflunomide for the treatment of relapsing-remitting MS between 2003 and 2020.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2003-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who developed skin cancer | From Index drug dispensation to the first of the following events, whichever occurred first: development of skin cancer; lost to follow-up; death; administrative end of follow-up; initiation of a comparator drug, assessed up to 180 months.
  In this outcome measure, participants who developed skin cancer after receiving the respective DMT treatments are reported. ICD 9/10 codes were used for the diagnosis of skin cancer (melanoma and non-melanoma skin cancers). Skin cancers were treated as a composite outcome of basal cell carcinoma, squamous cell carcinoma, and melanoma, as well as disaggregated by skin cancer subtypes.
Time to development of skin cancer | From Index drug dispensation to the first of the following events, whichever occurred first: development of skin cancer; lost to follow-up; death; administrative end of follow-up; initiation of a comparator drug, assessed up to 180 months.
  Time to development of skin cancer is defined as the time from the index date (drug initiation) to the development of skin cancer. ICD 9/10 codes were used for the diagnosis of skin cancer (melanoma and non-melanoma skin cancers). Skin cancers were treated as a composite outcome of basal cell carcinoma, squamous cell carcinoma, and melanoma, as well as disaggregated by skin cancer subtypes.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jia A, Kuramoto L, Khakban A, Sio WS, Traboulsee A, De Vera MA, Oh J, Loree J, Tam R, Lynd LD, Cragg JJ. Fingolimod and risk of skin cancer among individuals with multiple sclerosis: a population-based cohort study protocol. BMJ Open. 2025 Jan 23;15(1):e088924. doi: 10.1136/bmjopen-2024-088924. PMID 39855661